CLINICAL TRIAL: NCT02795546
Title: Effect of Alendronate With β - TCP Bone Substitute in Surgical Therapy of Periodontal Intra-osseous Defects: A Randomized, Controlled Clinical Trial.
Brief Title: Effect of Alendronate With β - TCP Bone Substitute in Surgical Therapy of Periodontal Intra-osseous Defects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Rohini Naineni, MDS, Reader, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMVIDS/PER/0029/2014
Record Dates: First submitted 2016-05-31; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Intrabony Periodontal Defect
Keywords: periodontal regeneration
MeSH Terms: interventions — Alendronate; beta-tricalcium phosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): 400µg Alendronate sodium+ β-TCP + saline. 400µg alendronate sodium is combined with beta-tricalcium phosphate bone substitute and wetted with saline and used as bone grafting material in periodontal intra-osseous defects.
  Interventions: Drug: Alendronate sodium; Biological: beta-tricalcium phosphate bone substitute
- Control group (Active Comparator): β-TCP + saline Beta-tricalcium phosphate bone substitute and wetted with saline and used as bone grafting material in periodontal intra-osseous defects.
  Interventions: Biological: beta-tricalcium phosphate bone substitute

INTERVENTIONS:
Drug: Alendronate sodium — 400µg of alendronate sodium is combined with beta-tricalcium phosphate bone graft and implanted in periodontal intra-osseous defects as a single, local dose.
  Other Names: fossamax, osteofos
  Arms: Test group
Biological: beta-tricalcium phosphate bone substitute — beta-tricalcium phosphate bone graft is implanted in periodontal intra-osseous defects.
  Other Names: cerasorb, sorbone

SUMMARY:
The aim of the present study was to evaluate the bone formation potential of 400µg alendronate delivered in β-TCP in the treatment of periodontal intra-osseous defects.

DETAILED DESCRIPTION:
The aim of the present study was to evaluate the bone formation potential of 400µg alendronate(ALN) delivered in β-TCP in the treatment of periodontal intra-osseous defects.

Materials and Methods: Thirty patients with periodontal defects were randomly assigned to 400µg ALN + β-TCP + saline (test) group and β-TCP + saline (active-control) group. Clinical parameters like clinical attachment level (CAL) gain, probing depth (PD) reduction, post-operative gingival recession (GR) were assessed from the baseline, 3 months and 6 months recordings. Radiographic parameters like linear bone growth (LBG), percentage bone fill (%BF), change in alveolar crest height (ACH) were assessed from baseline and 6 months radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients having an intra-osseous defect with probing depth ≥ 7mm at baseline, presence of a ≥ 4mm vertical inter-proximal bone defect with at least one bony wall after surgical debridement and with no history of previous periodontal therapy were included into the study

Exclusion Criteria:

* Patients with known systemic diseases, aggressive periodontitis, smoking habit, known or suspected allergy to bisphosphonates, pregnant and lactating women, study tooth exhibiting tooth mobility greater than grade II and class III furcation defect were excluded from the study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Linear bone growth | change from baseline and 6 months
  Linear bone growth (LBG) was calculated as the difference between the cemento-enamel junction(CEJ) to base of defect (BD) distance at baseline and CEJ to BD distance at 6 months in radiographs.

SECONDARY OUTCOMES:
clinical attachment level (CAL) | change from baseline and 6 months
  distance between the cemento-enamel junction and base of the pocket

IPD SHARING:
Plan to Share IPD: No
statistical data will be provided.

REFERENCES:
- [Result] Gupta J, Gill AS, Sikri P. Evaluation of the relative efficacy of an alloplast used alone and in conjunction with an osteoclast inhibitor in the treatment of human periodontal infrabony defects: a clinical and radiological study. Indian J Dent Res. 2011 Mar-Apr;22(2):225-31. doi: 10.4103/0970-9290.84292. PMID 21891890
- [Result] Sharma A, Pradeep AR. Clinical efficacy of 1% alendronate gel as a local drug delivery system in the treatment of chronic periodontitis: a randomized, controlled clinical trial. J Periodontol. 2012 Jan;83(1):11-8. doi: 10.1902/jop.2011.110091. Epub 2011 May 4. PMID 21542734
- [Result] Veena HR, Prasad D. Evaluation of an aminobisphosphonate (alendronate) in the management of periodontal osseous defects. J Indian Soc Periodontol. 2010 Jan;14(1):40-5. doi: 10.4103/0972-124X.65438. PMID 20922078